CLINICAL TRIAL: NCT03417544
Title: A Phase II Study of Atezolizumab in Combination With Pertuzumab Plus High-dose Trastuzumab for the Treatment of Central Nervous System Metastases in Patients With Her2-positive Breast Cancer
Brief Title: Atezolizumab + Pertuzumab + Trastuzumab In CNS Mets In BC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nancy Lin, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Nancy Lin, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-546
Record Dates: First submitted 2018-01-16; First posted 2018-01-31 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: HER2-positive Metastatic Breast Cancer; Central Nervous System Metastases
Keywords: HER2-positive metastatic Breast Cancer; Central Nervous System Metastases
MeSH Terms: interventions — atezolizumab; pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB (Experimental): Patients will receive the following treatment:
  * Atezolizumab (IV) every 3 weeks (q3w)]
  * Pertuzumab (loading dose ), followed q3w thereafter by a predetermined dose in the protocol via IV)
  * High-dose Trastuzumab weekly for the first 24 weeks, and thereafter trastuzumab q3w).
  Interventions: Drug: ATEZOLIZUMAB; Drug: PERTUZUMAB; Drug: TRASTUZUMAB

INTERVENTIONS:
Drug: ATEZOLIZUMAB — (IV) every 3 weeks
  Other Names: Tecentriq
Drug: PERTUZUMAB — Loading dose, followed every 3 weeks thereafter by a predetermined dose in the protocol via IV
  Other Names: Perjeta
Drug: TRASTUZUMAB — Predetermined dose per protocol via IV, weekly for 24 weeks and after every 3 weeks
  Other Names: Herceptin

SUMMARY:
This research study is studying a drug called atezolizumab as a possible treatment HER2-positive metastatic breast cancer (MBC) that has spread to the brain.

The names of the study drugs involved in this study are:

* Atezolizumab
* Pertuzumab
* Trastuzumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied. It also means that the FDA (U.S. Food and Drug Administration) has not approved the combination of atezolizumab, trastuzumab, and pertuzumab for use in humans. The FDA has not approved atezolizumab for this specific disease but it has been approved for other uses.

* Atezolizumab is a protein that affects the immune system by blocking the PD-L1 pathway. The PD-L1 pathway controls the body's natural immune response, but for some types of cancer the immune system does not work as it should and is prevented from attacking tumors. Atezolizumab works by blocking the PD-L1 pathway, which may help the immune system identify and catch tumor cells.
* Pertuzumab and trastuzumab are targeted therapies approved by the FDA to be used alone or in combination with a chemotherapy drug to treat HER2-positive metastatic breast cancer that hasn't been treated with either trastuzumab or chemotherapy yet.
* Pertuzumab and trastuzumab are called "targeted therapies" because they work by attaching themselves to specific receptors on the surface of breast cancer cells, known as HER2 receptors. When these targeted therapies attach to HER2 receptors, the signals that tell the cells to grow are blocked and the cancer cell may be marked for destruction by your immune system. This process allows pertuzumab and trastuzumab to help slow or stop the growth of the breast cancer. Pertuzumab and trastuzumab target different areas of the HER2 cell, so they are believed to work together more effectively.

In this research study, investigators are looking to see how well the cancer responds to the combination of atezolizumab in combination with pertuzumab and trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

- Eligibility will be assessed as part of the screening procedures for all patients.

* Pathologically confirmed HER2-positive MBC by local laboratory with the following requirements: HER2 overexpressed or amplified (immunohistochemistry of 3+ or HER2 gene amplification by in situ hybridization with a ratio of HER2-gene signals to centromere 17 signals ≥ 2.0 or average HER2 copy number ≥ 6.0 signals/cells).
* At least one measurable CNS metastasis, defined as ≥ 10 mm in at least one dimension
* Unequivocal evidence of new and/or progressive brain metastases, and at least one of the following scenarios:

  * Treated with SRS or surgery with residual un-treated lesions remaining. Such participants are eligible for immediate enrollment on this study providing that at least one untreated lesion is measurable
  * Participants who have had prior WBRT and/or SRS and then whose lesions have subsequently progressed are also eligible. In this case, lesions which have been treated with SRS may be considered as target lesions if there is unequivocal evidence, in the opinion of the treating physician, of progression following SRS.
  * Participants who have not previously been treated with cranial radiation (e.g., WBRT or SRS) are eligible to enter the study, but such participants must be asymptomatic from their CNS metastases and not requiring corticosteroids for symptom control.
  * Both participants who present with systemic stable/absent or progressive disease are eligible to this trial, as long as they fulfill one of the above criteria.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Left ventricular ejection fraction (LVEF) ≥ 50% by echocardiogram (echo) or multigated acquisition (MUGA) scan within 28 days before day 1 of study.
* Stable dose of dexamethasone 2mg or less for at least 7 days prior to initiation of treatment
* Concurrent administration of other anti-cancer therapy during the course of this study is not allowed. Note that concurrent use of supportive care medications (e.g. anti-resorptive agents, pain medications) is allowed.
* The subject is 18 years old.
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,000/μl
  * platelets ≥75,000/μl
  * hemoglobin ≥9 g/dL
  * total bilirubin ≤1.5mg/dL (upper limit of normal) except subject with documented Gilbert's syndrome (≤5 x ULN) or liver metastasis, who must have a baseline total bilirubin ≤3.0 mg/dL;
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN ≤ 5.0 × institutional ULN for patients with documented liver metastases.
  * albumin >2.5mg/dL
  * serum creatinine ≤ 1.5 mg/dL (or glomerular filtration rate ≥ 60 ml/min as determined by the Cockcroft-Gault equation)
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 8 days of initiating protocol therapy.
* The effects of atezolizumab on the developing human fetus are unknown and radiotherapy has known teratogenic effects so women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and 4 months after completion of atezolizumab administration.
* The subject is capable of understanding and complying with the protocol and has signed the informed consent document.

Exclusion Criteria:

* Visceral crisis or impending visceral crisis at time of screening.
* CNS complications for whom urgent neurosurgical intervention is indicated (e.g., resection, shunt placement).
* Known leptomeningeal or brainstem metastases [Defined as positive CSF cytology and/or unequivocal radiological evidence of clinically significant leptomeningeal involvement. CSF sampling is not required in the absence of suggestive symptoms to exclude leptomeningeal involvement].
* Treatment with high dose systemic corticosteroids defined as dexamethasone > 2mg/day or bioequivalent within 7 days of initiating therapy.
* Patients unable to undergo gadolinium contrast-enhanced MRI or receive IV contrast for any reason (e.g., due to pacemaker, ferromagnetic implants, claustrophobia, extreme obesity, hypersensitivity).
* Chemotherapy or targeted therapy within 14 days prior to cycle 1 day 1 of protocol therapy.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* No washout is required for endocrine therapy. If a patient has been on endocrine therapy within 28 days of study entry, that same endocrine therapy is permitted to be continued during protocol therapy, at the investigator's discretion, as is continuation of ovarian suppression in premenopausal women. Starting a new endocrine therapy during protocol therapy is not permitted
* Current use or history of receiving a non-approved, investigational treatment within 14 days prior to cycle 1 day 1 of protocol therapy
* Subjects with a history of hypersensitivity to compounds of similar biologic composition to atezolizumab or any constituent of the product
* The subject has an uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, congestive heart failure-New York Heart Association Class III or IV, active ischemic heart disease, myocardial infarction within the previous six months, uncontrolled diabetes mellitus, gastric or duodenal ulceration diagnosed within the previous 6 months, chronic liver or renal disease, or severe malnutrition.
* The subject is pregnant or breast-feeding
* No active, second potentially life-threatening cancer
* Has had major surgery within 21 days before cycle 1, day 1
* Active infection requiring iv antibiotics at day 1 of cycle 1
* Participant has a medical condition that requires chronic systemic steroid therapy or on any other form of immunosuppressive medication. For example, patients with autoimmune disease that requires systemic steroids or immunosuppression agents should be excluded. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs, resulting in dyspnea at rest
* The participant is known to be positive for the human immunodeficiency virus (HIV), HepBsAg, or HCV RNA. HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with atezolizumab.
* Has received a live vaccine within 28 days of planned start of study therapy.
* Known intolerance to trastuzumab or pertuzumab or atezolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB: Patients will receive the following treatment:
  * Atezolizumab (IV) every 3 weeks (q3w)]
  * Pertuzumab (loading dose ), followed q3w thereafter by a predetermined dose in the protocol via IV)
  * High-dose Trastuzumab weekly for the first 24 weeks, and thereafter trastuzumab q3w).
  ATEZOLIZUMAB: (IV) every 3 weeks
  PERTUZUMAB: Loading dose, followed every 3 weeks thereafter by a predetermined dose in the protocol via IV
  TRASTUZUMAB: Predetermined dose per protocol via IV, weekly for 24 weeks and after every 3 weeks
Period: Overall Study
Arm/Group | ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 50 [35 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
ECOG PS [Count of Participants; unit: Participants] — ECOG PS stands for Eastern Cooperative Oncology Group Performance Status, which is a scale used to assess how a patient's disease is progressing and how it affects their daily living abilities. The score is discrete and in the range of 0 to 5, higher score indicates worse patient performance.
  Participants
    0 | 12
    1 | 7
Stage at Initial Diagnosis [Count of Participants; unit: Participants] — The clinical stage at initial diagnosis in breast cancer is typically described using the TNM staging system, which takes into account the size of the primary tumor (T), whether the cancer has spread to nearby lymph nodes (N), and whether it has metastasized (spread to distant organs or tissues) (M). The stage is described as Roman numerals from 0 to IV, with higher numbers indicating a more advanced stage of cancer.
  Participants
    I | 1
    II | 5
    III | 5
    IV | 5
    Not IV, but otherwise unknown | 3
Hormone Receptor Status of Primary Tumor [Count of Participants; unit: Participants] — The Hormone Receptor Status of a primary breast tumor is defined using estrogen receptor (ER) and progesterone receptor (PR) status. HR-positive tumors were defined as having either ER-positive and/or PR-positive cells, while HR-negative tumors were defined as having neither ER-positive nor PR-positive cells.
  Participants
    ER and PR positive | 7
    ER positive/PR negative | 2
    ER negative/PR positive | 1
    ER and PR negative | 9
Hormone Receptor Status of Metastatic Tumor [Count of Participants; unit: Participants] — The Hormone Receptor Status of Metastatic Tumor is defined using estrogen receptor (ER) and progesterone receptor (PR) status. HR-positive tumors were defined as having either ER-positive and/or PR-positive cells, while HR-negative tumors were defined as having neither ER-positive nor PR-positive cells.
  Participants
    ER and PR positive | 1
    ER positive/PR negative | 2
    ER negative/PR positive | 1
    ER and PR negative | 10
    Unknown | 5
HER-2 Status of Primary Tumor (IHC) [Count of Participants; unit: Participants] — HER-2, also known as human epidermal growth factor receptor 2, is a protein that promotes the growth of cancer cells. The primary tumor was HER-2 positive by immunohistochemistry (IHC), indicating overexpression of the HER-2 protein. The primary tumor was HER-2 negative by immunohistochemistry (IHC), indicating no or low expression of the HER-2 protein.
  Participants
    Negative (0,1+) | 2
    Equivocal (2+) | 0
    Positive (3+) | 13
    Not Done | 4
HER-2 Status of Primary Tumor (FISH) [Count of Participants; unit: Participants] — HER-2 status of a primary breast tumor can also be determined using fluorescence in situ hybridization (FISH), which is another laboratory test that provides information about the HER-2 gene. The primary tumor was HER-2 positive by FISH, indicating amplification of the HER-2 gene. The primary tumor was HER-2 negative by FISH, indicating no amplification of the HER-2 gene.
  Participants
    Equivocal (4<= copy number <6 and HER2/CEP17 ratio <2.0) | 1
    Positive (copy number >=6 or HER2/CEP17 ratio >=2.0) | 8
    Not Done | 10
Measurable Disease by RECIST 1.1 [Count of Participants; unit: Participants]
  Yes | 7
  No | 12
Tissue Available at Baseline [Count of Participants; unit: Participants]
  Yes | 17
  No | 2
Sites of Disease at Study Entry [Count of Participants; unit: Participants]
  Breast or chest wall | 18
  Other | 1
Lines of Chemotherapy for Metastasis or Recurrence [Count of Participants; unit: Participants]
  None | 1
  1 line | 4
  2 lines | 6
  > 2 lines | 8
Use of Corticosteroids [Count of Participants; unit: Participants]
  Yes | 5
  No | 14
Prior Brain Surgery [Count of Participants; unit: Participants]
  Yes | 6
  No | 13

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Overall Response Rate in CNS
Description: The proportion of patients who had confirmed complete response or confirmed partial response, assessed using neuro-oncology-brain metastases (RANO-BM) criteria. RANO-BM assess the response of brain metastases to treatment, using MRI scan. There are four categories as results: Complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD), which is separately defined as disappearance of all target lesions, at least a 30% decrease in the sum of the diameters of target lesions, neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as progressive disease (PD) and at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest) or the appearance of one or more new lesions.
Time Frame: Participants were evaluated for response every 6 weeks for the first 24 weeks and then every 9 weeks thereafter, through study completion, an average of 24 weeks in the real study data
Measure: Count of Participants; unit: Participants
Arm/Group | ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB
Number analyzed (Participants) | 19
Participants | 2

2. Secondary Outcome: Objective Non-CNS Response Rates
Description: The proportion of patients who had confirmed complete response or partial response, according to response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria. RECIST is used to assess the response of solid tumors to treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB
Number analyzed (Participants) | 19
Participants | 1

3. Secondary Outcome: Clinical Benefit Rate in CNS at 18 Weeks
Description: The proportion of patients who had stable disease, confirmed partial response or complete response, respectively, >=18 weeks, according to RANO-BM criteria
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB
Number analyzed (Participants) | 19
Participants | 8

4. Secondary Outcome: Patient Reported Outcomes by MDASI-BT Stratified by CBR at 18 Weeks
Description: Evaluated by M.D. Anderson Symptom Inventory Brain Tumor (MDASI-BT). MDASI-BT assess 13 symptom items and 6 interference items from the core MDAST as well as 9 symptoms specific to brain tumors, and generate Symptom Severity Score (SSS) and Symptom Interference Score (SIS) separately. The scale of the scores are in a range of 0 to 10, where 0 represents "not present" or "not severe," and 10 represents "as bad as you can imagine" or "most severe." A higher score indicates a higher level of symptom severity.
  Mean of the scores are reported across groups with and without CBR at 18 weeks and in baseline, week 9 and week 24.
Time Frame: 24 weeks
Population: We only report the SSS and SIS scores that are available and stratified by with or without CBR at 18 weeks, thus the sample size in different categories differ from the overall sample size
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB
Number analyzed (Participants) | 18
score on a scale
  SSS Score for patients with CBR at 18 weeks at Baseline: number analyzed (Participants) | 7
  SSS Score for patients with CBR at 18 weeks at Baseline | 1.8 (1.2)
  SSS Score for patients with CBR at 18 weeks at Week 9: number analyzed (Participants) | 7
  SSS Score for patients with CBR at 18 weeks at Week 9 | 1.5 (0.9)
  SSS Score for patients with CBR at 18 weeks at Week 24: number analyzed (Participants) | 6
  SSS Score for patients with CBR at 18 weeks at Week 24 | 1.7 (1.3)
  SSS Score for patients without CBR at 18 weeks at Baseline: number analyzed (Participants) | 11
  SSS Score for patients without CBR at 18 weeks at Baseline | 1.9 (1.2)
  SSS Score for patients without CBR at 18 weeks at Week 9: number analyzed (Participants) | 8
  SSS Score for patients without CBR at 18 weeks at Week 9 | 1.9 (1.1)
  SSS Score for patients without CBR at 18 weeks at Week 24: number analyzed (Participants) | 10
  SSS Score for patients without CBR at 18 weeks at Week 24 | 2.5 (1.4)
  SIS Score for patients with CBR at 18 weeks at Baseline: number analyzed (Participants) | 7
  SIS Score for patients with CBR at 18 weeks at Baseline | 4.0 (2.3)
  SIS Score for patients with CBR at 18 weeks at Week 9: number analyzed (Participants) | 7
  SIS Score for patients with CBR at 18 weeks at Week 9 | 2.8 (2.6)
  SIS Score for patients with CBR at 18 weeks at Week 24: number analyzed (Participants) | 6
  SIS Score for patients with CBR at 18 weeks at Week 24 | 2.6 (3.4)
  SIS Score for patients without CBR at 18 weeks at Baseline: number analyzed (Participants) | 11
  SIS Score for patients without CBR at 18 weeks at Baseline | 2.2 (2.1)
  SIS Score for patients without CBR at 18 weeks at Week 9: number analyzed (Participants) | 8
  SIS Score for patients without CBR at 18 weeks at Week 9 | 2.4 (2.4)
  SIS Score for patients without CBR at 18 weeks at Week 24: number analyzed (Participants) | 10
  SIS Score for patients without CBR at 18 weeks at Week 24 | 4.2 (2.9)

5. Secondary Outcome: Patient Reported Outcomes by EQ-5D Stratified by CBR at 18 Weeks
Description: Evaluated by EuroQol Five Dimension Questionnaire (EQ-5D) evaluations assessments to assess the general health status of patients enrolled in the study. EQ-5D scores are assessed with five dimensions with the range of 0 to 5, and a higher score indicates worse health.
  Mean of the scores are reported across groups with and without CBR at 18 weeks and in baseline, week 9 and week 24.
Time Frame: 24 weeks
Population: We only report the EQ-5D scores that are available and stratified by with or without CBR at 18 weeks, thus the sample size in different categories differ from the overall sample size
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB
Number analyzed (Participants) | 18
units on a scale
  Patients with CBR at 18 weeks at Baseline: number analyzed (Participants) | 7
  Patients with CBR at 18 weeks at Baseline | 0.7 (0.5)
  Patients with CBR at 18 weeks at Week 9: number analyzed (Participants) | 8
  Patients with CBR at 18 weeks at Week 9 | 0.5 (0.4)
  Patients with CBR at 18 weeks at Week 24: number analyzed (Participants) | 6
  Patients with CBR at 18 weeks at Week 24 | 0.7 (0.9)
  Patients without CBR at 18 weeks at Baseline: number analyzed (Participants) | 11
  Patients without CBR at 18 weeks at Baseline | 0.9 (0.7)
  Patients without CBR at 18 weeks at Week 9: number analyzed (Participants) | 8
  Patients without CBR at 18 weeks at Week 9 | 0.8 (0.4)
  Patients without CBR at 18 weeks at Week 24: number analyzed (Participants) | 10
  Patients without CBR at 18 weeks at Week 24 | 1.4 (0.7)

6. Secondary Outcome: Investigator-Assessed Neurological Evaluation (NANO) Stratified by CBR at 18 Weeks
Description: Evaluated by physician assessed Neurological Assessment in Neuro-Oncology (NANO) scale. The NANO scale is a quantifiable evaluation of 9 relevant neurologic domains based on direct observation and testing conducted during visits. The score defines overall response criteria and is with the range of 0 to 4. Higher score means worse response to the treatment.
  Mean of the scores are reported across groups with and without CBR at 18 weeks and in baseline, week 9 and week 24.
Time Frame: 24 weeks
Population: We only report the NANO scores that are available and stratified by with or without CBR at 18 weeks, thus the sample size in different categories differ from the overall sample size
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB
Number analyzed (Participants) | 18
units on a scale
  Patients with CBR at 18 weeks at Baseline: number analyzed (Participants) | 8
  Patients with CBR at 18 weeks at Baseline | 0.03 (0.08)
  Patients with CBR at 18 weeks at Week 9: number analyzed (Participants) | 8
  Patients with CBR at 18 weeks at Week 9 | 0.1 (0.13)
  Patients with CBR at 18 weeks at Week 24: number analyzed (Participants) | 5
  Patients with CBR at 18 weeks at Week 24 | 0.17 (0.27)
  Patients without CBR at 18 weeks at Baseline: number analyzed (Participants) | 10
  Patients without CBR at 18 weeks at Baseline | 0.1 (0.14)
  Patients without CBR at 18 weeks at Week 9: number analyzed (Participants) | 10
  Patients without CBR at 18 weeks at Week 9 | 0.18 (0.24)
  Patients without CBR at 18 weeks at Week 24: number analyzed (Participants) | 9
  Patients without CBR at 18 weeks at Week 24 | 0.39 (0.27)

7. Secondary Outcome: Clinical Benefit Rate in CNS at 24 Weeks
Description: The proportion of patients who had stable disease, confirmed partial response or complete response, respectively, >=24 weeks, according to RANO-BM criteria
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB
Number analyzed (Participants) | 19
Participants | 6

ADVERSE EVENTS:
Time Frame: All adverse events were reported after initiation of study treatment and until 30 days after the last dose of study treatment or until initiation of new systemic anti-cancer therapy, an average of one and a half years
Description: Serious Adverse Events are defined as any events with grade 3 or higher. Other Adverse Events include any grade 1 and 2 events and those exceed 5% frequency threshold are reported.
Arm/Group | ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB
All-Cause Mortality (participants affected / at risk) | 1/19
Serious Adverse Events (participants affected / at risk) | 10/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB (N=19)
Anemia (Blood and lymphatic system disorders) | 3
Heart failure (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Other (General disorders) | 1
Fatigue (General disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
Weight loss (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Edema cerebral (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ATEZOLIZUMAB, PERTUZUMAB, TRASTUZUMAB (N=19)
Anemia (Blood and lymphatic system disorders) | 5
Lymph node pain (Blood and lymphatic system disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 2
Sinus tachycardia (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 5
Blurred vision (Eye disorders) | 2
Dry eye (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 2
Optic nerve disorder (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Fecal incontinence (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 16
Fever (General disorders) | 2
Gait disturbance (General disorders) | 5
Malaise (General disorders) | 1
Pain (General disorders) | 6
Immune system disorders - Other, specify (Immune system disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Papulopustular rash (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 5
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 7
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 3
Weight gain (Investigations) | 4
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Ataxia (Nervous system disorders) | 5
Cognitive disturbance (Nervous system disorders) | 3
Concentration impairment (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 4
Dysarthria (Nervous system disorders) | 1
Dysesthesia (Nervous system disorders) | 2
Facial muscle weakness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 11
Memory impairment (Nervous system disorders) | 4
Nervous system disorders - Other, specify (Nervous system disorders) | 2
Paresthesia (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 4
Seizure (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Spasticity (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 3
Anxiety (Psychiatric disorders) | 5
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 4
Mania (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Urine discoloration (Renal and urinary disorders) | 1
Dyspareunia (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 1
Lymphedema (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT03417544/Prot_SAP_000.pdf